CLINICAL TRIAL: NCT00872534
Title: A Randomized, Single-Blind, Endoscopic Evaluation Of Upper GI Mucosal Damage Induced By PL-2200 Versus Aspirin In Healthy Volunteers
Brief Title: Endoscopic Evaluation of Upper Gastrointestinal (GI) Mucosal Damage Induced by PL-2200 Versus Aspirin in Healthy Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PLx Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PL-ASA-002
Record Dates: First submitted 2009-03-10; First posted 2009-03-31 (Estimated); Results first posted 2015-08-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Upper Gastrointestinal Mucosal Damage
Keywords: To evaluate the acute gastrointestinal safety of PL-2100.
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- PL-2200 (Experimental): PL-2200 is an NSAID product containing 325mg of acetylsalicylic acid and phosphatidylcholine in a neutral lipid matrix.
  Interventions: Drug: acetylsalicylic acid
- Aspirin (Active Comparator): Immediate release 325mg aspirin
  Interventions: Drug: acetylsalicylic acid

INTERVENTIONS:
Drug: acetylsalicylic acid — 325mg once a day for 7 days

SUMMARY:
To determine the gastrointestinal safety of PL-2200 versus immediate-release aspirin by assessing endoscopic gastroduodenal mucosal injury at approved daily cardiac-protective doses of aspirin (325 mg) in normal healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥50 to ≤75 years of age.
* Subject is healthy.
* Subject has a BMI between 20 and 32
* If female and of child bearing potential, subject has a negative pregnancy test and is not nursing.

Exclusion Criteria:

* Subject has abnormal screening/baseline laboratory parameters or endoscopic observations deemed clinically significant by the Investigator.
* Subject has an active Helicobacter pylori infection.
* Subject has a prior GI ulcer, bleeding, obstruction or perforation.
* Subject has taken aspirin or any aspirin containing product within the last 4 weeks, or a non-aspirin NSAID product within 2 weeks.
* Subject has taken any of the following medications within 2 weeks prior to enrollment: Any anti-platelet agents, anti-coagulants or selective serotonin reuptake inhibitors.
* Subject has used an investigational agent within the past 30 days.
* Subject has hypersensitivity or contraindications to aspirin, ibuprofen, or other NSAID.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2009-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Byron L Cryer, MD, Principal Investigator — Dallas VA; Frank L Lanza, MD, Principal Investigator — Houston Institute for Clinical Research; Michael E Schwartz, DO, Principal Investigator — Jupiter Research; Alan J Kivitz, MD, Principal Investigator — Altoona Arthritis and Osteoporosis Center; Phillip B Miner, MD, Principal Investigator — Oklahoma Foundation for Digestive Research; Howard Schwartz, MD, Principal Investigator — Miami Research Associates
Locations (6):
- United States (6):
  - Jupiter Research, Jupiter, Florida
  - Miami Research Associates, South Miami, Florida
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Altoona Arthritis and Osteoporosis Center, Altoona, Pennsylvania
  - Dallas VA Medical Center, Dallas, Texas
  - Houston Center For Clinical Research, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PL-2200 | Aspirin
Started | 100 | 104
Completed | 97 | 101
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PL-2200 | Aspirin | Total
Number analyzed (Participants) | 100 | 104 | 204
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (6.35) | 56.6 (6.00) | 57.3 (6.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 56 | 60 | 116

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Subjects With Gastroduodenal Erosions and Ulcers.
Description: Incidence of subjects with gastroduodenal composite scores of 3 or 4 (> 5 erosions or 1 or more ulcers 3 mm or greater in length with unequivocal depth).
Time Frame: After 7 days of study medication
Measure: Number; unit: participants
Arm/Group | PL-2200 | Aspirin
Number analyzed (Participants) | 91 | 90
participants
  Gastroduodenal Composite Score of 3 or 4 (NO) | 72 | 54
  Gastroduodenal Composite Score of 3 or 4 (YES) | 19 | 36

ADVERSE EVENTS:
Arm/Group | PL-2200 | Aspirin
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/104
Other Adverse Events (participants affected / at risk) | 8/100 | 14/104
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PL-2200 (N=100) | Aspirin (N=104)
Nausea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Stomach Ulcer (Gastrointestinal disorders) | 3 (3) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Standard Confidentiality Agreement